CLINICAL TRIAL: NCT04921852
Title: The Comparation of Lateral Sagittal Infraclavicular and Costoclavicular Approach in Brachial Plexus Blocks
Brief Title: The Comparation of Lateral Sagittal Infraclavicular and Costoclavicular Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Suleymank, medical doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: costoclavicular
Record Dates: First submitted 2021-05-30; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Upper Extremity Problem
Keywords: costoclavicular block; Lateral sagittal Infraclavicular block; brachial plexus block; block onset time

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- costoclavicular group (Active Comparator)
  Interventions: Procedure: costoclavicular brachial plexus block
- lateral sagittal group (Active Comparator)
  Interventions: Procedure: lateral sagittal infraclavicular block

INTERVENTIONS:
Procedure: costoclavicular brachial plexus block — A transverse scan with an portable USG machine with a high-frequency linear array transducer ((Logiq E, General Electric, ABD) will be performed immediately below the midpoint of the clavicle and over the medial infraclavicular fossa. 20 ml of a mixture of 0.25% bupivacaine, 1% lidocaine will be injected in to the middle of the three brachial plexus cords with an echogenic SonoTAP(Pajunk GmbH Medizintechnologie, Geisingen, Germany) block needle under USG guidance .Readiness for surgery time will be evaluated after costoclavicular block.
  Arms: costoclavicular group
Procedure: lateral sagittal infraclavicular block — A sagittal scan with an portable USG machine with a high-frequency linear array transducer ((Logiq E, General Electric, ABD) will be performed medial to the coracoid process to obtain a transverse view of the axillary artery.20 ml of a mixture of 0.25% bupivacaine, 1% lidocaine will be injected posterior to the axillary artery near to the three cords of brachial plexus with an echogenic SonoTAP(Pajunk GmbH Medizintechnologie, Geisingen, Germany) block needle under USG guidance.Readiness for surgery time will be evaluated after lateral sagittal infraclavicular block.
  Arms: lateral sagittal group

SUMMARY:
In this study, the investigators aimed to compare the block dynamics and characteristics of the two approaches while providing effective analgesia and safe anesthesia of the Ultrasound-guided Lateral sagittal Infraclavicular and costoclavicular approach in Brachial plexus blocks.

DETAILED DESCRIPTION:
Participants between the ages of 18-70 with the American Society of Anesthesiology (ASA) score I-II-III will be included in the study. All participants will be evaluated preoperatively and information will be given about the anesthetic method to be applied. Demographic data and ASA scores of the participants will be recorded.

All of the participants included in the study will be taken to the regional anesthesia application room in the operating room approximately 1 hour before the operation. After standard anesthesia monitoring (electrocardiography, pulsoximetry, non-invasive blood pressure), all participants will be given an iv vascular access with a 20 or 22 G cannula from the arm that will not be operated.

All blocks will be made using portable US machine and echogenic block needle.

For all blocks, 20 ml of a mixture of 0.25% bupivacaine, 1% lidocaine will be used.

An overall (average) sensory and motor score was also calculated for every participants and at each time point assessed by averaging the VRS sensory or motor scores of all the 4 nerves will be tested preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 to 3
* 18-70 age
* hand , wrist , forearm and elbow surgery

Exclusion Criteria:

* refusal to participate,
* pregnancy,
* body mass index of 30 kg/m2 or greater
* history of allergy to local anesthetic drugs
* prior surgery over the infraclavicular fossa,
* preexisting neurological deficit
* coagulopathy
* infection over infraclavicular fossa.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-06-07 (Estimated); Primary Completion 2021-09-07 (Estimated); Study Completion 2021-10-07 (Estimated)

PRIMARY OUTCOMES:
readiness for surgery time | 30 minute
  Sensory block, defined as a loss of sensation to cold (ice), in the cutaneous distribution of the median (MN), radial (RN), ulnar (UN), and musculocutaneous (MCN) nerves will be assessed and graded according to a VRS (0-100, 100 = normal sensation and 0 = no sensation). Motor blockade of each of the 4 nerves in the ipsilateral upper extremity was also assessed and graded according to a 3-point qualitative scale (2 = normal motor power, 1 = paresis, and 0 = paralysis).Onset of sensory and motor blockade for each nerve was defined as the time (onset time) it took to achieve a sensory VRS of 30 or less and motor power grade of 1 or less, respectively.Time to readiness for surgery was defined as the time it took to achieve an overall sensory score of 30 or less and motor power grade of 1 or less, in all the 4 nerves tested.

SECONDARY OUTCOMES:
block performance time | 5 minute
  the time it took from the start of the local skin infiltration to the end of the local anesthetic injection

IPD SHARING:
Plan to Share IPD: No